CLINICAL TRIAL: NCT02516254
Title: Comparison of the Efficacy of Vitamin D-fortified Bread Versus Vitamin D Supplement in Healthy Adults: a Randomized Controlled Clinical Trial
Brief Title: Assessment of the Efficacy of Vitamin D-fortified Bread in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, Ph.D., Professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 054-574
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: vitamin D; fortified bread; efficacy; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fortified bread (Experimental): daily intake of fortified bread (1000IU vitamin D per 50 g) plus placebo
  Interventions: Dietary Supplement: fortified bread
- supplement (Experimental): daily intake of plain bread (50 g) plus supplement (1000 IU per tablet)
  Interventions: Dietary Supplement: supplement
- placebo (Placebo Comparator): daily intake of plain bread plus placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: fortified bread — 50 g of fortified bread + placebo daily
  Other Names: FB
  Arms: fortified bread
Dietary Supplement: supplement — vitamin D supplement+ plain bread
  Other Names: SP
  Arms: supplement
Dietary Supplement: placebo — plain bread+placebo
  Other Names: PP
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of daily intake of fortified bread with vitamin D on serum 25-hydroxyvitamin D level, glycemic and lipidemic status in healthy subjects compared to vitamin D supplement.

DETAILED DESCRIPTION:
Sixty apparently healthy subjects will be selected. Participants who are receiving vitamin D, calcium or omega-3 supplements within the last three months will be excluded. Subjects will be assigned randomly to one of the three intervention groups: 1.fortified bread+placebo,2. plain bread+vitamin D supplements,3. plain bread+placebo. Each participant will consume 50 g of bread and supplement or placebo every day for 2 months.

At the first and last visits, dietary and laboratory assessments will be performed for all subjects. Primary outcomes are improvement in vitamin D status and secondary outcome is improvement of glycemic and lipidemic markers and prevention of problems related to hypovitaminosis D.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 50 years
* healthy subjects
* no receiving vitamin D or omega-3 supplement in past 3 months

Exclusion Criteria:

* receiving vitamin D or omega-3 supplement during the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D (nmol/L) | 8 weeks

SECONDARY OUTCOMES:
serum glucose (mg/dL) | 8 weeks
serum triglyceride (mg/dL) | 8 weeks
serum total cholesterol (mg/dL) | 8 weeks
serum LDL | 8 weeks
serum HDL (mg/dL) | 8 weeks
serum PTH (pg/mL) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, PhD, Study Chair — Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran